## **Artificial Intelligence Detection of Bladder Tumors under Endoscopy**

## **Informed Consent Form**

Version: 1.0

Date: 2023-11-15

| Name: | Gender: | Age: |
|-------------|--------------|------|
| Department: | Patient No.: | |

## Informed Consent Form for Surgical Video Collection, Intraoperative Photography, and Clinical Data Collection

Dear Patient,

Thank you for your trust in our hospital, and we wish you a quick recovery.

All the clinical researches are based on the collection of clinical data, medical photos, surgical videos, and many types of medical data.

We hope to obtain your consent to collect your personal demographic information, medical records, laboratory test data, imaging, photographs, and surgical videos during your diagnosis and treatment process. These data will be used for clinical diagnosis and treatment, teaching, and medical research purposes. When the research results are published or reported, we will hide all your personal information to protect your privacy from being compromised. Your personal information will not be disclosed to other irrelevant individuals unless with your permission. To ensure that the researches are conducted in accordance with regulations and to guarantee that your rights are not compromised, members from government or ethics review committee may review your medical data as necessary.

You have the right not to sign this informed consent form, and you also have the right to withdraw your signed consent form at any time. Whether you agree or not will

| not affect your diagnosis and treatment, nor will it affect your relationship with | tne |
|---|---|
| medical staff. The doctor has illustrated the above content to me, and I confirm that I under the confirm the confirm that I under the confirm that I under the confirm that I under the confirm th | erstand |
| the content above completely. After careful consideration, I agree to provide my demographic information, medical records, laboratory test data, imaging, photographic and surgical videos and other medical data for clinical, teaching, and medical repurposes. | y persor<br>graphs, |
| Signature of Patient or Authorized Representative: | |
| Signature Date: | |
| Signature of Doctor: | |
| Signature Date: | |